CLINICAL TRIAL: NCT03752684
Title: Oxalobacter Formigenes Colonization and Oxalate Excretion in Healthy Adults
Brief Title: Oxalobacter Formigenes Colonization and Urinary Oxalate Excretion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, John Knight, Associate Professor, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: IRB-131212001; R01DK087967 (NIH)
Record Dates: First submitted 2018-10-22; First posted 2018-11-26 (Actual); Results first posted 2025-06-10 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Calcium Oxalate Urolithiasis
Keywords: Oxalobacter formigenes; oxalate; kidney stones
MeSH Terms: conditions — Nephrolithiasis, Calcium Oxalate; Kidney Calculi

STUDY DESIGN:
Intervention Model Description: Evaluate urinary oxalate excretion before and after colonization with the oxalate degrading bacterium Oxalobacter formigenes
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Colonization with Oxalobacter formigenes (Experimental): Subjects not colonized with Oxalobacter formigenes will be equilibrated to a moderately high oxalate/ low calcium oxalate controlled diet and collect 24-hour urines to measure oxalate excretion Subjects will then be colonized with Oxalobacter formigenes(Intervention). Following colonization with Oxalobacter formigenes, urinary oxalate will be measured to determine the impact of colonization on the same controlled diet
  Interventions: Dietary Supplement: Moderately high oxalate/low calcium diet non-colonized; Dietary Supplement: Oxalobacter formigenes; Dietary Supplement: Moderately high oxalate/low calcium diet colonized

INTERVENTIONS:
Dietary Supplement: Moderately high oxalate/low calcium diet non-colonized — Subjects will be instructed to ingest a controlled diet moderately high in oxalate before colonization
Dietary Supplement: Oxalobacter formigenes — Subjects will ingest live preparation of O. formigenes
Dietary Supplement: Moderately high oxalate/low calcium diet colonized — Subjects will be instructed to ingest a controlled diet moderately high in oxalate after colonization

SUMMARY:
The purpose of this research study is to assess the efficacy of ingesting a small amount of the harmless bacterium Oxalobacter formigenes in establishing residence in the guts of healthy participants and to determine whether this influences the oxalate passed in urine.

DETAILED DESCRIPTION:
Adults that are not colonized with O. formigenes, have no history of stone disease, and are in good health as judged by their medical history and a complete metabolic profile of their serum, will be recruited from within the greater Birmingham area.

Participants not colonized with O. formigenes will consume a controlled diet containing moderately high levels of oxalate (210-240 mg per day), and low levels of calcium (500 - 700 mg per day) and collect 24-hour urines to measure oxalate excretion. Following completion of urine collections, participants will ingest live O.formigenes and one week later stool will be provided to test for colonization with O.formigenes. Participants that are successfully colonized with O.formigenes will then repeat 24 hour urine collections on the same high oxalate, low calcium diet. Controlled diets will be prepared in the Metabolic Kitchen of the UAB Clinical Research Unit (CRU). Sustainability of colonization will be determined over time. Loss of colonization will be confirmed by having the subject consume an oxalate-rich meal with subsequent testing for O. formigenes.

ELIGIBILITY:
Inclusion Criteria:

* Good health as judged from a medical history and reported medications
* Not colonized with O. formigenes

Exclusion Criteria:

* History of any hepatic, renal, bowel or endocrine disease or any other condition that may influence the absorption, transport or urinary excretion of ions, which will compromise the interpretation of results
* colonized with O. formigenes
* abnormal urine chemistries or blood metabolic profiles

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2018-04-02 (Actual); Primary Completion 2023-04-27 (Actual); Study Completion 2025-05-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Knight, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited within the Greater Birmingham area
Groups:
- Colonization With Oxalobacter Formigenes: Moderately high oxalate/low calcium diet non-colonized: Participants not colonized with O. formigenes will be instructed to ingest the controlled diet and collect 24-hour urines to measure oxalate excretion
  Oxalobacter formigenes: Participants will then ingest a live preparation of O. formigenes
  Moderately high oxalate/low calcium diet colonized: Participants successfully colonized with O. formigenes will be instructed to ingest the same controlled diet consumed prior to colonization
Period: Overall Study
Arm/Group | Colonization With Oxalobacter Formigenes
Started | 26
Completed | 22
Not Completed | 4
Not completed — Lost to Follow-up | 4

BASELINE CHARACTERISTICS:
Groups:
- Colonization With Oxalobacter Formigenes: Moderately high oxalate/low calcium diet non-colonized: Participants not colonized with O.formigenes will collect 24-hour urines on the controlled diet
  Oxalobacter formigenes: Participants will ingest live preparation of O. formigenes
  Moderately high oxalate/low calcium diet colonized: Participants successfully colonized with O.formigenes will collect 24-hour urines on the same controlled diet
Arm/Group | Colonization With Oxalobacter Formigenes
Number analyzed (Participants) | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 22
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 8
  White | 13
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 22
Body Mass Index [Mean (Standard Deviation); unit: kg per m2] | 29 (5)

OUTCOME MEASURES:

1. Primary Outcome: Percent Decrease in Urinary Oxalate Excretion After Colonization With O.Formigenes
Description: Mean 24-hour urine oxalate excretion after colonization with O.formigenes was compared with mean 24-hour urine oxalate before colonization
Time Frame: 4 days
Measure: Mean (Full Range); unit: Percentage decrease in urinary oxalate
Groups:
- Colonization With Oxalobacter Formigenes: Moderately high oxalate/low calcium diet non-colonized: Participants not colonized with O.formigenes will collect 24 urines on the controlled diet
  Oxalobacter formigenes: Participants will ingest live preparation of O. formigenes
  Moderately high oxalate/low calcium diet colonized: Participants successfully colonized with O.formigenes will collect 24 urines on the controlled diet
Arm/Group | Colonization With Oxalobacter Formigenes
Number analyzed (Participants) | 22
Percentage decrease in urinary oxalate | 14 [-12 to 46]

2. Secondary Outcome: Percentage Decrease in Stool Oxalate Content After Colonization With O.Formigenes
Description: Mean stool oxalate content after colonization with O.formigenes was compared with mean stool oxalate before colonization
Time Frame: 4 days
Measure: Mean (Full Range); unit: Percentage decrease in stool oxalate
Groups:
- Colonization With Oxalobacter Formigenes: Moderately high oxalate/low calcium diet non-colonized: Participants not colonized with O.formigenes collected stool on the controlled diet
  Oxalobacter formigenes: Participants ingested live preparation of O. formigenes
  Moderately high oxalate/low calcium diet colonized: Participants successfully colonized with O.formigenes collected stool on the controlled diet
Arm/Group | Colonization With Oxalobacter Formigenes
Number analyzed (Participants) | 22
Percentage decrease in stool oxalate | 54 [1 to 93]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for 4 weeks after ingestion of O.formigenes
Arm/Group | Colonization With Oxalobacter Formigenes
All-Cause Mortality (participants affected / at risk) | 0/22
Serious Adverse Events (participants affected / at risk) | 0/22
Other Adverse Events (participants affected / at risk) | 0/22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-05-22): https://cdn.clinicaltrials.gov/large-docs/84/NCT03752684/Prot_SAP_000.pdf
  • Informed Consent Form (2021-01-06): https://cdn.clinicaltrials.gov/large-docs/84/NCT03752684/ICF_001.pdf